CLINICAL TRIAL: NCT05370820
Title: Prevention of Postpartum Hemorrhage: Pharmacokinetics (PK) Abd Pharmacodynamics (PD) of Tranexamic Acid
Brief Title: Prevention of Postpartum Hemorrhage With Tranexamic Acid
Acronym: Optimum OB-TXA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: George Washington University (Other); University of Maryland (Other); University of North Carolina (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Homa Ahmadzia, MD, MD, PI, Inova Health Care Services
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: INOVA-2024-39; R01HD110109 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-05-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cesarean Delivery (Experimental)
  Interventions: Drug: Tranexamic acid; Other: No intervention
- Vaginal Delivery (Experimental)
  Interventions: Drug: Tranexamic acid; Other: No intervention
- Morbidly Obese (Experimental)
  Interventions: Drug: Tranexamic acid; Other: No intervention
- No TXA (No Intervention)

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic Acid 1000 mg administered intravenously via infusion over 10 minutes.
  Arms: Cesarean Delivery; Morbidly Obese; Vaginal Delivery
Drug: Tranexamic acid — Tranexamic Acid 1000 mg administered intravenously via push over 2 minutes.
  Arms: Cesarean Delivery; Morbidly Obese; Vaginal Delivery
Drug: Tranexamic acid — Tranexamic Acid 1000 mg administered intramuscularly.
  Arms: Cesarean Delivery; Morbidly Obese; Vaginal Delivery
Other: No intervention — Control group with no administration of Tranexamic Acid.
  Arms: Cesarean Delivery; Morbidly Obese; Vaginal Delivery

SUMMARY:
In part 1 of the study, the investigators conducted a prospective, open-label, dose finding pharmacokinetic (PK) study in 43 pregnant 3rd trimester women scheduled for non-emergent cesarean section.

The investigators administered three doses of the drug (5 mg/kg, 10 mg/kg and 15 mg/kg) in an escalating fashion by cohort with the lowest dose first. The drug was administered intravenously at the time of umbilical cord clamping for a non-emergent cesarean section. A maximum of 1 gram was administered. TXA serum levels at several time points after delivery were assayed to see if they reach the target plasma concentration of 10 microg/mL. A PK model was constructed for determining the optimal TXA dose administered at parturition.

In part 2 of the study, the investigators aim to compare PKPD endpoints using prophylactic TXA via IV and IM routes administered pre-cord clamp. The investigators will administer 1000 mg TXA within 10 minutes of skin incision via intravenous infusion (up to n=15), intravenous bolus < 2 minutes (up to n=15) and intramuscular injection (up to n=15). The investigators will target women undergoing scheduled cesarean delivery greater than 34 weeks gestation, women undergoing vaginal delivery > 34 weeks of gestation and morbidly obese women (BMI>=40) undergoing either a vaginal or cesarean delivery. The investigators will use advanced modeling techniques to determine time to achieve PKPD targets and duration remaining at those targets. The goal will be to determine how the optimal dose may vary if route of administration is modified. The investigators plan to enroll 45 patients in addition to the 43 that were enrolled during part 1. Our goal is to 30 participants, but the investigators will enroll 45 to account for lost to follow-up. The investigatorsalso aim to enroll 30 patients undergoing vaginal delivery and 30 morbidly obese women (BMI > 50) undergoing either a vaginal or cesarean delivery but the investigators will enroll 45 patients for each of these groups to account for loss to follow up. In addition, the investigators will enroll 30 pregnant patients receiving no medication acting as the control group, but the investigators will enroll 45 to account for loss to follow up.

DETAILED DESCRIPTION:
The study will enroll 45 additional third trimester pregnant women scheduled for nonemergent cesarean sections who are at high risk for hemorrhage. The investigators plan to enroll 30, but to account for lost to follow-up, the investigators will enroll 45. The investigators will also enroll 30 pregnant patients > 34 weeks of gestation undergoing vaginal delivery, and 30 morbidly obese (BMI >= 40) pregnant patients undergoing either vaginal or cesarean delivery. However, the investigators will enroll 45 patients in each of these two groups to account for loss to follow up. The investigators will also enroll 45 patients as a control group that will not receive TXA. The total number of enrolled patients will thus be 223.

A total of 1 gram of TXA will be administered to patients prior to fetal delivery via three different routes of administration: IV infusion, IV push, and IM injection. The subjects in each group will be divided into three subgroups:

Group 1: Up to 15 subjects, TXA dose: 1 gram, Route: IV infusion over 10 minutes Group 2: Up to 15 subjects, TXA dose: 1 gram, Route: IV Push for <2 minutes Group 3: Up to 15 subjects, TXA dose: 1 gram, Route: IM Injection

Plasma sampling: Timing of samples will be relative to the end of drug administration (t = 0) and include: Pre-drug administration, 5-10 minutes, 30-60 minutes, 60-90 minutes, 1.5-3 hours, 3-4 hours, 4-5 hours, 7-8 hours, and 10-18 hours. Each volume of blood draw will be approximately 7-9 mL. Actual times of plasma sampling will be documented. A second IV will be required for participating in the study. Citrated plasma samples will be centrifuged and supernatant will be stored at -70 degree Celsius. Breast milk sampling of no more than 2 mL per time point will occur at time points coinciding with maternal feedings.

ELIGIBILITY:
Inclusion Criteria:

* Women who are scheduled to under medically indicated cesarean section at greater than 34+0 weeks gestation or women who are scheduled to undergo an elective cesarean section at 39+0 weeks gestation in accordance with recommendations from the American Congress of Obstetricians and Gynecologists
* Women who are indicated to have a vaginal delivery at > 34+0 weeks gestation.
* Pregnant women with normal serum creatinine (serum creatinine < 0.9) within 2 weeks of estimated/scheduled delivery
* Women between the ages of 18 and 50 years old
* Ability to understand and the willingness to sign a written informed consent form and HIPAA Authorization.

Exclusion Criteria:

* active thrombotic or thromboembolic disease
* a history of arterial or venous thromboembolic event
* inherited thrombophilia or preexisting conditions that predisposes them to thromboembolic events (i.e. lupus, antiphospholipid syndrome, thrombocytosis or thrombophilic thrombocytopathy)
* a subarachnoid hemorrhage
* acquired defective color vision
* history of seizure disorder
* known renal dysfunction (serum creatinine = or >0.9)
* multiple gestations (twin or triplet pregnancies)
* hypersensitivity to Tranexamic acid or anti-fibrinolytic therapy
* history of liver dysfunction at the discretion of the investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
LI30 (Fibrinolysis Marker) | T(0) to 1 day postpartum
  Change in LI30 (lysis index at 30 minutes) as measured by ROTEM, before and after TXA injection, to assess the pharmacodynamic effects of TXA.

CONTACTS AND LOCATIONS:
Overall Officials: Homa K Ahmadzia, MD, Principal Investigator — Inova Health Care Services
Locations (2):
- United States (2):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Undecided